CLINICAL TRIAL: NCT04974086
Title: Feasibility and Acceptability of an Electronic Clinical Decision Support Tool for Adolescent Sexual and Reproductive Health Services
Brief Title: Electronic Sexual Reproductive Health CDS Tool at the Children's Hospital of Philadelphia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-018609; K23MH119976 (NIH)
Record Dates: First submitted 2021-04-21; First posted 2021-07-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sexual and Reproductive Health
MeSH Terms: conditions — Coitus | interventions — Compact Disks; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Single arm prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDS Tool Evaluation (Experimental): All participants will receive intervention and feasibility, acceptability, and usability of intervention will be assessed from each participant cohort group.
  Interventions: Other: Sexually transmitted infection (STI) testing clinical decision support (CDS) tool

INTERVENTIONS:
Other: Sexually transmitted infection (STI) testing clinical decision support (CDS) tool — The intervention, called the STI Testing CDS tool, includes integrating STI testing guideline prompts into the electronic health record (EHR). The prompt guides clinicians to assess and broadly respond to adolescents' sexual health behaviors through EHR survey data. Through the CDS tool, clinicians will be prompted to provide comprehensive and evidence-based sexual health care for teens including, for example: providing patient-facing education about sexual preventative health topics and facilitating ordering of HIV and sexually transmitted infection (STI) laboratory tests to improve both risk-based and routine annual preventative screening.

SUMMARY:
Many studies show early detection of sexual activity in adolescents can improve their health management and that primary care pediatricians would benefit from supports to address adolescent health, including sexual and reproductive health. The primary objective of this study is to develop and evaluate the feasibility, acceptability, and usability of a sexually transmitted infection (STI) testing clinical decision support (CDS) tool within the electronic health record (EHR) among clinicians, adolescent patients, and their parents. Secondary objectives include assessment of the CDS tool's impact on clinical measures. The STI Testing CDS tool will be embedded within clinical practice and evaluated through a single-armed prospective cohort study of primary care clinicians, adolescent patients, and parents. The STI Testing CDS tool that will support pediatric clinicians by providing evidence-based sexual health-related screening, treatment, and referrals, as needed.

DETAILED DESCRIPTION:
The STI Testing CDS tool will be embedded within the electronic health record (EHR) and will be evaluated to include feasibility (through medical record review for EHR utilization data), pediatric clinician acceptability and usability of the intervention (using surveys and semi-structured interviews), and adolescent and parent acceptability of the approach (using surveys). The secondary outcomes include measures of clinical impact, including ordering (and the results) of gonorrhea, chlamydia, and HIV screening labs.

Three cohorts of participants will be involved in the study: 1) Clinicians (attending physicians, nurse practitioners, and pediatric residents), 2) their English-speaking adolescent patients, and 3) their parents at included primary care sites.

The first 100 adolescent patients for whom the CDS tool is used will be approached in-person or remotely via text message or phone call after the clinical visit to complete a brief survey on the acceptability of the treatment provided at the visit, acceptability of that treatment, satisfaction with potential treatment outcomes, and if they engaged in any conversations with their parent(s) about any treatment provided at the visit.

Similarly, parents of those first 100 adolescent patients will be approached in-person or remotely via text message or phone call after the clinical visit to complete a brief survey on the acceptability of the approach to adolescent care workflow (not any specifics about the actual care provided) as well as any conversations about the visit that occurred between the parent and adolescent after the visit. Contact information, including phone number, for potential adolescent and parent participants will be retrieved from the adolescent's medical record. Additionally, Investigators will approach 50 pediatric clinicians in-person or remotely via email to complete a brief survey and semi-structured interview on the feasibility, acceptability, and usability of the CDS tool. Pediatric clinicians are eligible if they care for adolescent patients and have used the STI Testing CDS tool in practice.

Results from clinician surveys and semi-structured interviews will ensure that the CDS tool design meets clinicians' needs - ensuring a level of usability, functionality, and usefulness that supports pediatric clinicians' delivery of sexual and reproductive health care services to adolescents.

Secondary outcome measures aimed at assessing the clinical impact of the STI Testing CDS tool will include:

* Number of gonorrhea, chlamydia, and HIV tests ordered as a result of the CDS tool,
* And, the number of positive gonorrhea, chlamydia, and HIV tests ordered as a result of the CDS tool.

This study presents no more than minimal risk to study participants, as this is a study aimed to assess the creation of a tool that helps to improve upon the current delivery of sexual and reproductive health services provided through pediatric primary care.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients who meet the following inclusion criteria will be eligible: Sexually transmitted infection (STI) testing clinical decision support (CDS) tool is used at the preventive care visit, age 13 years or older, English-speaking
* Parents who meet the following inclusion criteria will be eligible: Attend a preventive care visit with their adolescent child, are 18 years of age or older, English-speaking, have a smartphone, personal contact information is available in their child's electronic health record (EHR)
* Clinicians who meet the following inclusion criteria will be eligible: Use the STI Testing CDS tool at a preventative care visit with an adolescent patient

Exclusion Criteria:

• Subjects who do not meet the above inclusion criteria will be excluded.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-02-11 (Actual)

PRIMARY OUTCOMES:
Usability of a sexually transmitted infection (STI) testing clinical decision support (CDS) tool among clinicians as assessed by the SUS. | 1 day
  The System Usability Scale (SUS) is a validated 10-item tool used for measuring subjective assessments of usability. This survey will be presented to pediatric clinicians using the sexual reproductive health (SRH) CDS tool and they will be asked to rate how much they agree/disagree with 10 statements related to the tool's usability.
Acceptability of a sexually transmitted infection (STI) testing clinical decision support (CDS) tool among clinicians as assessed through qualitative interviews. | 1 day
  Qualitative interviews will be conducted with pediatric clinicians who use the CDS tool. This interview will be one-on-one and ask questions that assess attitudes towards using the tool and feedback on how to improve the tool.
Feasibility of a sexually transmitted infection (STI) testing clinical decision support (CDS) tool among clinicians as assessed through qualitative interviews. | 1 day
  Qualitative interviews will be conducted with pediatric clinicians who use the CDS tool. This interview will be one-on-one and ask questions that assess feasibility of consistently using the tool in practice and feedback on how to improve use of the tool within the adolescent encounter.
Acceptability of a sexually transmitted infection (STI) testing clinical decision support (CDS) tool among adolescents | 1 day
  This will be measured through a survey for adolescents who presented for a well child care visit and completed the Adolescent Health Questionnaire (a health screener used as standard care in all well child care visits). The survey consists of 36 potential questions about acceptability of a questionnaire part of standard well visits and of potential reproductive health services they received during their visit, attitudes towards privacy of their visit and discussions with their provider, & feedback on discussions that occurred between them and a parent/guardian after their visit.
Acceptability of a sexually transmitted infection (STI) testing clinical decision support (CDS) tool among parents of adolescents | 1 day
  This will be measured through a survey for parents of adolescents who were present during their child's well child care visit. The survey consists of 22 potential questions about acceptability of a questionnaire that includes measuring perspectives on sexual healthcare for teens as part of standard well care, acceptability of their child receiving confidential services part of standard well care, & feedback on discussions that occurred between them and their child after their visit.

SECONDARY OUTCOMES:
Assessment of the CDS tool's impact on the number of sexually transmitted infection/human immunodeficiency virus (STI/HIV) tests ordered. | up to 2 years
  This will be measured by the difference in pre- and post-intervention metrics for the number of gonorrhea, chlamydia, and HIV tests ordered as a result of the CDS tool. These metrics will be measured by pre- and post-intervention data analytics provided by the Children's Hospital of Philadelphia (CHOP) Department of Biomedical and Health Informatics (DBHI).
Assessment of the CDS tool's impact on the number of positive STI/HIV tests. | up to 2 years
  This will be measured by the difference in pre- and post-intervention metrics for the number of positive STI/HIV tests as a result of the CDS tool. These metrics will be measured by pre- and post-intervention data analytics provided by the Children's Hospital of Philadelphia (CHOP) Department of Biomedical and Health Informatics (DBHI).

CONTACTS AND LOCATIONS:
Overall Officials: Brian P. Jenssen, MD, Principal Investigator — Primary care pediatrician and researcher
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No